CLINICAL TRIAL: NCT06230276
Title: How do the Currently Available HCL Systems Manage Missed Meal Bolus? The Comparison of Glycemic Outcomes After Missed Meal Bolus Between MiniMed 780G, Tandem Control-IQ and Ypsomed CamAPS
Brief Title: Managing of Missed Meal Bolus by HCL Systems
Acronym: NOELLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zdeněk Šumník (Other)
Responsible Party: Sponsor-Investigator, Zdeněk Šumník, Head of the Department of Pediatrics, University Hospital, Motol
Organization: University Hospital, Motol (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1B_23N01
Record Dates: First submitted 2023-12-17; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Enteral Nutrition; Breakfast

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention with and without premeal bolus (Experimental)
  Interventions: Other: enteral nutrition (Resource Fibre, 2 kcal/ml) for breakfast

INTERVENTIONS:
Other: enteral nutrition (Resource Fibre, 2 kcal/ml) for breakfast — Participants who are already treated by one of the HCL systems (MiniMed 780G, Tandem Control-IQ, Ypsomed CamAPS) will have a precisely defined amount of enteral nutrition (Resource Fibre, 2 kcal/ml) for breakfast during eight different days under predetermined conditions. They will administer premeal bolus only for half of these meals.

SUMMARY:
The goal of this interventional study is to compare glycemic outcomes after missed meal bolus in children and adolescents with type 1 diabetes (CwD) treated by one of the three most common used types of hybrid closed loop (HCL) systems - Medtronic MiniMed 780G, Tandem Control-IQ, Ypsomed CamAPS. The main questions it aims to answer are:

* Do the glycemic outcomes (area under the curve of glucose concentration change, maximal glucose rise from baseline, time to maximal glucose rise from baseline, CGM parameters) vary after missed meal bolus among different types of HCL systems?
* Does the type of insulin analog influence glycemic outcomes after a missed meal bolus?

Participants will have a precisely defined amount of enteral nutrition (Resource Fibre, 2 kcal/ml) for breakfast during eight different days under predetermined conditions. They will administer premeal bolus only for half of these meals.

ELIGIBILITY:
Inclusion Criteria:

* children with type 1 diabetes (CwD) 9.00-18.99 years old
* use of continuous glucose monitoring (CGM) >70% of the time 14 days before a regular check-up in the outpatient clinic
* HCL use (MiniMed 780G, Tandem Control-IQ or Ypsomed CamAPS) >3 months
* duration of T1D >2 years
* baseline HbA1c level <58 mmol/mol (7.5%)
* weight > 30 kilograms
* without any medication influencing glycemia (f.e. gliflozins, systemic corticosteroids…)
* signed informed consent form with the study

Ages: 9 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Difference in an area under the curve of a glucose concentration change 4 hours after a meal (30 g and 50 g of carbohydrates) with a missed premeal bolus between individual HCL systems. | 4 hour after a meal

SECONDARY OUTCOMES:
Difference in a maximal glucose rise from baseline after a meal (30 g and 50 g of carbohydrates) with a missed premeal bolus between individual HCL systems. | 4 hours after a meal
Difference in time to maximal glucose rise from baseline after a meal (30 g and 50 g of carbohydrates) with a missed premeal bolus between individual HCL systems. | 4 hours after a meal
Difference in CGM parameters 4 hours after a meal (30 g and 50 g of carbohydrates) with a missed premeal bolus between individual HCL systems. | 4 hours after a meal
  time in range TIR (3.9-10.0 mmol/L; 70-180 mg/dL) time above range level 1 TAR1 (10.1-13.9 mmol/L; 181-250 mg/dL) time above range level 2 TAR2 (> 13.9 mmol/L; >250 mg/dL) time below range level 1 TBR1 (3.0-3.8 mmol/L; 54-69 mg/dL) time below range level 2 TBR2 (< 3.0 mmol/L; <54 mg/dL) time in tight range TITR (3.9-7.8 mmol/L; 70-140 mg/dL)
Difference in an area under the curve of a glucose concentration change 4 hours after a meal (30 g and 50 g of carbohydrates) with a missed premeal bolus between individual HCL systems using different types of insulin analogs | 4 hours after a meal
  insulin analogs - aspart and ultra-rapid lispro
Difference in a maximal glucose rise from baseline after a meal (30 g and 50 g of carbohydrates) with a missed premeal bolus between individual HCL systems using two different types of insulin analogs | 4 hours after a meal
  insulin analogs - aspart and ultra-rapid lispro
Difference in time to maximal glucose rise from baseline after a meal (30 g and 50 g of carbohydrates) with a missed premeal bolus between individual HCL systems using two different types of insulin analogs | 4 hours after a meal
  insulin analogs - aspart and ultra-rapid lispro
Difference in CGM parameters after a meal (30 g and 50 g of carbohydrates) with a missed premeal bolus between individual HCL systems using insulin ultra-rapid lispro | 4 hours after a meal
  time in range TIR (3.9-10.0 mmol/L; 70-180 mg/dL) time above range level 1 TAR1 (10.1-13.9 mmol/L; 181-250 mg/dL) time above range level 2 TAR2 (> 13.9 mmol/L; >250 mg/dL) time below range level 1 TBR1 (3.0-3.8 mmol/L; 54-69 mg/dL) time below range level 2 TBR2 (< 3.0 mmol/L; <54 mg/dL) time in tight range TITR (3.9-7.8 mmol/L; 70-140 mg/dL)
Difference in CGM parameters after a meal (30 g and 50 g of carbohydrates) with a missed premeal bolus between individual HCL systems using insulin aspart. | 4 hours after a meal
  time in range TIR (3.9-10.0 mmol/L; 70-180 mg/dL) time above range level 1 TAR1 (10.1-13.9 mmol/L; 181-250 mg/dL) time above range level 2 TAR2 (> 13.9 mmol/L; >250 mg/dL) time below range level 1 TBR1 (3.0-3.8 mmol/L; 54-69 mg/dL) time below range level 2 TBR2 (< 3.0 mmol/L; <54 mg/dL) time in tight range TITR (3.9-7.8 mmol/L; 70-140 mg/dL)

CONTACTS AND LOCATIONS:
Locations (1):
- Motol University Hospital, Prague, Czechia